CLINICAL TRIAL: NCT01189383
Title: IL15-DC Vaccine in Patients With High Risk Melanoma - Exploratory Phase I/II Trial
Brief Title: IL15 Dendritic Cell Vaccine for Patients With Resected Stage III (A, B or C) or Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 009-273; R01CA140602 (NIH)
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Malignant Melanoma Stage III; Malignant Melanoma Stage IV
Keywords: Melanoma; Vaccine; Dendritic Cell; Immune response; Safety; Efficacy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IL15-DC Vaccine (Experimental): Approximately 9 x 10^6 DCs will be injected (subcutaneously)total per vaccination visit. Patients will receive four vaccinations at weeks 0, 4, 8 and 12.At each scheduled vaccination the patient will receive a total of 3 injections, i.e., 3 mL injections at each of 3 anatomical locations.Injection sites are in upper and lower extremities. Subsequent DC injections will be rotated to different locations on the upper and lower extremities.
  Interventions: Biological: IL15-DC Vaccine

INTERVENTIONS:
Biological: IL15-DC Vaccine — Autologous dendritic cells manufactured with GM-CSF, IL15 and loaded with melanoma/HIV peptides and KLH; then activated with LPS and CD40 Ligand. Approximately 9 x 10^6 DCs will be injected (subcutaneously)total per vaccination visit. Patients will receive four vaccinations at weeks 0, 4, 8 and 12. At each scheduled vaccination the patient will receive a total of 3 injections, i.e., 3 mL injections at each of 3 anatomical locations.Injection sites are in upper and lower extremities. Subsequent DC injections will be rotated to different locations on the upper and lower extremities.

SUMMARY:
The purpose of the study is to gather data on feasibility as well as immune and clinical efficacy of of a dendritic cell vaccine using IL15 in patients with resected stage III or stage IV melanoma

DETAILED DESCRIPTION:
IL15 is a T cell growth factor that pre-clinical data overwhelmingly suggests could have a very important role in cancer immunotherapy. A desirable property for a dendritic cell vaccine directed against cancer is the ability to efficiently prime naïve, tumor associated antigen specific T cells into potent CTLs. Results of studies in healthy volunteers have shown that IL15 DCs are particularly efficient at priming functional melanoma specific CD8+ T cells. The use of IL15 in the manufacture of the DC vaccine could result in an improved immunotherapy product.

ELIGIBILITY:
Inclusion Criteria:

* HLA A201 + phenotype
* Biopsy-proven melanoma, Stages III (A, B and C) or stage IV.- no evidence of disease at study entry
* Age: 21-75 years
* ECOG performance status 0-1
* Adequate marrow function
* Adequate hepatic function
* Adequate renal function
* Written informed consent

Exclusion Criteria:

* Subjects with measureable non-resectable melanoma
* Subjects who have had chemotherapy less than 4 weeks before starting trial
* Subjects who received IFN-a or GM-CSF less than 4 weeks before starting trial
* Subjects who received IL2 less than 4 weeks before starting trial
* Subjects with a baseline LDH greater than 1.1 times the ULN
* Subjects who are HIV positive
* Female subjects who are pregnant
* Subjects who have received corticosteroids or other immunosuppressive agents less than 4 weeks before starting trial
* Subjects who have asthma and/or are on treatment for asthma
* Subjects with angina pectoris
* Subjects with congestive heart failure
* Subjects with history of autoimmune disease including lupus, rheumatoid arthritis or thyroiditis
* Subjects with active infections including viral hepatitis
* Subjects with a history of neoplastic disease othe than melanoma within the last 5 years
* History of neoplastic disease within the last 5 years except for carcinoma in situ of the cervix, superficial bladder cancer or basal/squamous cell carcinoma of the skin.
* Subjects who present with open wounds

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Immune response | 14 weeks

SECONDARY OUTCOMES:
Quality of elicited melanoma specific CD8+ T cells | 14 weeks
Breadth of melanoma specific immunity | 24 weeks
Longevity of melanoma specific CD8+ T cell immunity | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Fay, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

REFERENCES:
- See also: Click here for more information on this study: IL15-DC Vaccine in Patients With High Risk Melanoma - Exploratory Phase I/II Trial — http://www.baylorhealth.com/AdvancingMedicine/GetInvolved/Pages/BRI_Display.aspx?IRBNumber=IRB-009-273